CLINICAL TRIAL: NCT01581463
Title: Phase 1 Single-Dose Study of the Pharmacokinetics of Sustained-Release Liothyronine Sodium (T3) in Healthy Subjects
Brief Title: A Study of Sustained-Release Liothyronine Sodium (T3) in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ipe, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BCT303
Record Dates: First submitted 2012-04-18; First posted 2012-04-20 (Estimated); Last update posted 2012-08-06 (Estimated); Status verified 2012-08

CONDITIONS: Healthy
Keywords: pharmacokinetics of oral T3
MeSH Terms: interventions — Triiodothyronine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Liothyronine, Sodium (Active Comparator): Healthy adults.
  Interventions: Drug: Liothyronine, Sodium

INTERVENTIONS:
Drug: Liothyronine, Sodium — Single 100-microgram (2 X 50 microgram) dose.

SUMMARY:
Liothyronine is indicated for the treatment of primary hypothyroidism. Between 6 and 10 Million in the United States and 80 Million patients world-wide are hypothyroid, usually the result of autoimmune thyroiditis called Hashimoto's Disease. Hypothyroid symptoms result from low levels of thyroid hormones (T4 and T3) in the blood due to inadequate thyroid hormone production by the thyroid gland. Every tissue in the body is a thyroid hormone target and hypothyroid symptoms can be debilitating.

BCT303 utilizes Liothyronine, Sodium as the active ingredient, the same Liothyronine salt utilized as the active ingredient in currently marketed products.

The current "gold standard" for treatment of hypothyroidism are products containing Levothyroxine (T4). T4 is known to be a pro-hormone, converted to the more active hormone T3 by deiodinases in various tissues. Patients on Levothyroxine therapy alone are occasionally not euthyroid as measured by clinical presentation, a condition hypothesized to result from low levels of T3 from inadequate T4 to T3 conversion. In addition, the efficiency of conversion of T4 to T3 is variable and dependent on the patho-physiologic state of the patient.

BCT303 contains Liothyronine, Sodium as the active ingredient. This product has a patented formulation and granulation procedure that solves multiple clinical and stability problems associated with T3-based products. Thus, BCT303 is designed to have:

1. Increased shelf stability to ensure the maintenance of claimed dosage.
2. A sustained-release profile to minimize side effects associated with spikes in serum T3 levels.
3. Uniformity of dose between production batches and between tablets.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults
* Must be able to swallow tablets

Exclusion Criteria:

* Hypothyroid Disease
* Pregnant Females

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-04; Primary Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Serum Total T3 | Four Days.

CONTACTS AND LOCATIONS:
Locations (1):
- Georgetown University Hospital, Washington D.C., District of Columbia, United States